CLINICAL TRIAL: NCT04068571
Title: Innovative Partnership for Universal Health Coverage
Brief Title: Enhancing Universal Health Coverage and Maternal, Newborn and Child Health in Kenya Through Digital Innovations
Acronym: UHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: African Population and Health Research Center (Other)
Collaborators: Amsterdam Institute for Global Health and Development (Other); PharmAccess (Unknown)
Responsible Party: Principal Investigator, Amanuel Abajobir, Co-investigator, African Population and Health Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AfricanPHRC
Record Dates: First submitted 2019-07-31; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Universal Health Coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PUSH intervention sites (Active Comparator): Clusters with I-PUSH intervention
  Interventions: Behavioral: I-PUSH
- No I-PUSH intervention sites (No Intervention): Clusters with no I-PUSH intervention

INTERVENTIONS:
Behavioral: I-PUSH — Innovative partnership for universal and sustainable healthcare
  Arms: I-PUSH intervention sites

SUMMARY:
This study aims at providing insights into Universal Health Coverage and evaluates the impact of I-PUSH program on maternal healthcare utilization, financial protection and women's empowerment, as well as to evaluate the impact of the LEAP training tool on community health volunteers and women's health literacy including their knowledge, behavior and uptake of respective services.

DETAILED DESCRIPTION:
The study will use a three-pronged approach: year-long weekly Financial and Health Diaries, Baseline and Endline surveys, and qualitative interviews. The Diaries and the Surveys will be carried out in two Counties, Kakamega and Kisumu (Kenya). The qualitative interviews will be carried out in the two counties and in Nairobi as an additional county. The study will use a cluster randomized control trial design in Kakamega to evaluate the impact of I-PUSH program. In Kisumu, selected households will be followed-up to capture the health-seeking behavior, health insurance, and health expenditure pattern of households over time. The study will be initially for 17 months and will continue for three years subject to additional funding.

ELIGIBILITY:
Inclusion Criteria:

* Targets for the intervention

Exclusion Criteria:

* Non-targets for the intervention

Ages: 15 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Health Care Utilization | 17 months
  Financial and health diaries will be collected on a weekly basis throughout the indicated study period
Maternal, Newborn and Child Health outcomes through out the continuum of care | 17 months
  Questionnaire based survey questions will be used to measure these outcomes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abajobir A, Maina D, Wambui E, Sidze EM. Association between maternal mental health and early childhood development, nutrition, and common childhood illnesses in Khwisero subcounty, Kenya. PLoS One. 2025 Jan 17;20(1):e0317762. doi: 10.1371/journal.pone.0317762. eCollection 2025. PMID 39823401
- [Derived] Abajobir A, de Groot R, Wainaina C, Njeri A, Maina D, Njoki S, Mbaya N, Donfouet HPP, Pradhan M, Janssens W, Sidze EM. The impact of i-PUSH on maternal and child health care utilization, health outcomes, and financial protection: study protocol for a cluster randomized controlled trial based on financial and health diaries data. Trials. 2021 Sep 15;22(1):629. doi: 10.1186/s13063-021-05598-7. PMID 34526072